CLINICAL TRIAL: NCT00471705
Title: Phase 3 Open-label Study of Efficacy and Safety of Miltefosine or Thermotherapy vs Glucantime for Cutaneous Leishmaniasis in Colombia.
Brief Title: Efficacy and Safety of Miltefosine or Thermotherapy for Cutaneous Leishmaniasis in Colombia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Dirección de Sanidad del Ejército de Colombia (DISAN) (Unknown); Ministerio de Salud y Protección Social, Colombia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PECET-001
Record Dates: First submitted 2007-05-07; First posted 2007-05-10 (Estimated); Results first posted 2010-07-14 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2009-06

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Miltefosine; Leishmaniasis; Glucantime; Thermotherapy; Colombia
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis; Hyperthermia | interventions — miltefosine; Hyperthermia, Induced; Meglumine Antimoniate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Miltefosine (Experimental): Miltefosine 2.5 mg/Kg/day with a maximum dose of 150 mg PO day.
  Interventions: Drug: Miltefosine
- Glucantime® (Active Comparator): Glucantime® 20 mg /Kg /day for 20 days (intramuscular)
  Interventions: Drug: Glucantime®
- Thermotherapy (Experimental): One session of local heat using a thermotherapy device at 50 celsius degrees during 30 seconds.
  Interventions: Device: Thermotherapy

INTERVENTIONS:
Drug: Miltefosine — Miltefosine 2.5 mg/Kg/day with a maximum dose of 150 mg PO day.
  Other Names: Impavido®
  Arms: Miltefosine
Device: Thermotherapy — One session of local heat using a thermotherapy device at 50 celsius degrees during 30 seconds.
  Other Names: Thermomed
  Arms: Thermotherapy
Drug: Glucantime® — Glucantime® 20 mg /Kg /day for 20 days (intramuscular)
  Other Names: Glucantime® (meglumine antimoniate)
  Arms: Glucantime®

SUMMARY:
Cutaneous leishmaniasis (CL) is a worldwide disease, endemic in 88 countries, that has shown an increasing incidence the last two decades. It is estimated that in 2005, about of 20,000 new cases of CL were diagnosed in Colombia.

So far, pentavalent antimony compounds have been considered the treatment of choice with a percentage of cure of about 85%. However, the high efficacy of these drugs is counteracted by their adverse events and disadvantages. Previous studies have shown that miltefosine could be a potential alternative of treatment for CL.

The main objective of this study is to evaluate the efficacy and safety of miltefosine or thermotherapy for the treatment for CL. In this study the efficacy of oral treatment of miltefosine 150 mg/day for 28 days or a thermotherapy device used for one session at 50 celsius degrees during 30 seconds will be compared with the standard treatment of intramuscular injections of 20 mg/Kg/day of pentavalent antimonials (GlucantimeÒ) for 20 days in CL parasitologically proven patients.

This trial will be conducted according to the International approved GCP (Good Clinical Practice) guidelines.

DETAILED DESCRIPTION:
Evaluation of Efficacy and Safety of Miltefosine for Cutaneous Leishmaniasis in Colombia Leishmaniasis is taking dramatic dimensions in Colombia, due to its rapid expansion, reemergence (which has made Colombia became in the second South American country in levels of annual incidence) the appearance of new infection sources, the entrance of the vector to the homes, the urbanization of the disease, the higher population in risk of infection, the absence of adequate medications ( safe, non-expensive, easily available, with oral or topic route of administration) and the higher resistance to the only available medication for its treatment. It is estimated that in 2005 more than 20,000 new cases were diagnosed; 10,265 of them among the Colombian military forces personnel, but it is well known that in most of the rural areas the major proportion of cases are not diagnosed and the people cannot reach to an adequate treatment and they have to use empiric options.

On the other hand, the Program for Research and Control in tropical diseases (PECET) is working among Tropical Diseases Research/World Health Organization(TDR/WHO) in the evaluation of drugs and vaccines against Leishmaniasis; besides, PECET belongs to the TDR/WHO Clinical Monitors groups, TDR/WHO Data Management and participates in the Initiative for Public Health Products Development Doctorate among five Asiatic universities. The Ministry of Social Protection is aware of the need of new therapeutic alternatives for Leishmaniasis and has requested to PECET to conduct a controlled clinical trial to determinate the efficacy and safety of Miltefosine compared with Glucantime for the treatment of Cutaneous Leishmaniasis (CL) in Colombia, even though previous, no conclusive trials, conducted in Guatemala and Colombia, have demonstrated efficacy this could be an alternative of treatment for this country.

Thermomed is a battery-operated medical device that delivers precisely controlled localized current field radio frequency heat to selectively destroy certain diseased tissue. Radio frequency energy is directed through the handset to the applicator that is placed in direct contact with the lesion. (the applicator contains a thermocouple to continuously monitor and control temperature to within 50º Celsius. The thermomed has been used for research on treatment for cutaneous leishmaniasis, and recent clinical studies have shown not only clinical improvement, but also that therapy elicits an immune response to the disease. Through this trial we will try to perform a conclusive clinical evaluation about this drug.

In summary, with this project to conduct a clinical trial to determine the efficacy and safety of Miltefosine or thermotherapy compared with Glucantime for treatment of CL in Colombian patients.

Population CL in is a remerging disease in Colombia affecting civilian and military population as well, sharing the same epidemiologic characteristics.

The selected population will be composed from National Army of Colombia soldiers from CL endemic areas (Caquetá, Meta, Guaviare, Putumayo, Córdoba, Antioquia and Chocó).

Treatment:

In this phase III, randomized open trial, subjects meeting inclusion criteria of the trial will be randomly allocated into two groups according to a randomization list. One group will be treated with 150 mg/day of oral miltefosine for 28 days a second group will be treated with thermotherapy device used for one session at 50 celsius degrees during 30 seconds and a third group will be treated with intramuscular injections of 20 mg/kg/day Glucantime® for 20 days. A written instruction sheet will be given to each included patient, and the patient will be instructed to contact the research team on appearance of symptoms suggesting severe side effects (intractable diarrhea and/or vomiting, symptoms of liver, kidney or hematopoietic system dysfunction. Until six weeks after the termination of the treatment, any patient who received oral miltefosine or was treated with thermotherapy and has active lesion will be treated with intramuscular Glucantime® injections (20mg/kg/day for 20 days).

Study development Schedule of activities Screening (-2 or day 0): Protocol explanation, invitation to participate, inform consent signature, parasitological diagnosis (Direct test), laboratory tests (Complete hemogram, Ureic Nitrogen (BUN), creatinine, amylase, Glutamic-pyruvic transaminase(GTP or ALT), glutamic-oxaloacetic transaminase(GOT or AST)).

Inclusion (Visit 1): Randomization, sampling of Cultures, physical examination, vital signs measure, oral treatment initiation (Miltefosine for 28 days) or Glucantime® intramuscular application initiation (for the 20 subsequent days) or thermotherapy ( Local heat), patient's clinical record, CRF (Case Report Format) fulfilling, lesions picture taking.

Visit 2 (Middle of treatment): Laboratory tests (Complete hemogram, BUN, creatinine, amylase, GOT, GPT), physical examination, vital signs measure, CRF (Case Report Format) fulfilling, Lesions picture taking.

Visit 3 (End of treatment, +10 days): Laboratory tests (Complete hemogram, BUN, creatinine, amylase, GTP, GOT), physical examination, vital signs measure, CRF (Case Report Format) fulfilling, lesions picture taking, Evaluation of treatment efficacy.

Visit 4 (Six weeks after treatment, ± 15 days): Physical examination, Vital signs measure, CRF (Case Report Format) fulfilling, lesions picture taking, evaluation of treatment efficacy.

Visit 5 (Three months after treatment, ± 30 days): Physical examination, Vital signs measure, CRF (Case Report Format) fulfilling, lesions picture taking, evaluation of treatment efficacy.

Visit 6 (Six months after treatment, ± 40 days): Physical examination, Vital signs measure, CRF (Case Report Format) fulfilling, lesions picture taking, evaluation of treatment efficacy.

Procedures:

Physical examination A complete physical examination will be realized and vital signs will be measured.

Blood samples withdrawn

Blood samples will be withdrawn from the antecubital vein to perform the following analyses:

* Creatinine and Blood Urea Nitrogen.
* Alanine transaminase (ALT)
* Aspartate transaminase (AST)
* Pancreatic amylase.
* Complete hemogram.

Technique for the sampling of cultures The sample for the culture may be obtained by suctioning the ulcer active edge in a phosphate-buffered saline solution (PBS) with antibiotics (1000 IU of crystalline Penicillin per cc), before it is put in the culture medium.

A tuberculin syringe 0.5 cc of PBS solution with antibiotics is used in the suction technique. Previous asepsis of the ulcer with alcohol at 70%, a needle is introduced into the dermis and through rotating movements a small amount of tissue is macerated by the needle bevel during about a minute, after which it is suctioned into the syringe. The sample is deposited in aseptic conditions into a NNN (Novy-MacNeal-Nicole ) culture medium and incubated at 26°C during 4 weeks. The strains are identified by species using the monoclonal antibodies.

Toxicity

The grade of toxicity will be evaluated according the following parameters:

* Systemic: Fever, Headache.
* Gastrointestinal: Nausea, vomiting, oral discomfort.
* Cardiovascular: cardiac rhythm, hypertension, hypotension.
* Musculoskeletal: Arthralgia (joint pain) , myalgia,

During the treatment and the follow-up visits, the patients will be asked about adverse events. Each adverse event will be classified by the physician as serious or non-serious A serious adverse event should meet one or more of the following criteria:

* Death
* Life-threatening (i.e., immediate risk of death)
* In-patient hospitalization or prolongation of existing hospitalization
* Persistent or significant disability/incapacity The presence of a serious adverse event that puts the patient's life at risk and/or requires immediate medical or surgical procedure will call for the discontinuation of the treatment and the initiation of the pertinent medical management of the patients. The study staff will notify the Adverse IEC/IRB of the University of Antioquia of any serious adverse event within 24 hours of having knowledge of it.

A non-serious adverse event will be classified as follows:

Mild: The patients are aware of their symptoms and/or signs, but those are tolerable. They do not require medical intervention or specific treatment.

Moderate: Patients present troubles that interfere with their daily activities. They require medical intervention or specific treatment.

Severe: The patients are unable to work or to attend their daily activities. They require medical intervention or specific treatment.

The possible relationship between the adverse events and the tested medication will be classified by the investigator on the basis of his/her clinical judgment and the following definitions:

Definitely related: Event can be fully explained by the administration of the tested medication.

Probably related: Event is most likely to be explained by the administration of the tested medication rather than other medications or by the patient's clinical state.

Possibly related: Event may be explained by the administration of the tested medication or other medications or by the patient's clinical state.

Not related: Event is most likely to be explained by the patient's clinical state or other medications, rather than the tested one.

Data analysis phase. The healing rate will be calculated according to each group (treatment and control) by intention to treat and by protocol. Subgroups will be established depending on the clinical response, adverse events and according to Leishmania specie. Besides, the characteristics of the lesion (size, localization, type of lesion), demographic characteristics and how long the healing takes after the treatment is settled.

In all cases significance test will be performed to compare both treatments.

Endpoints Primary Clinical response: Complete re-epithelization of all lesions with disappearance of induration (with or without scar). No parasitological evaluation will be done on clinically cured lesions determined until 45 days posttreatment.

Clinical improvement: Reduction of a ≥50% area of induration and ulcer compared with immediately previous evaluation.

Secondary:

Treatment failure: No change or increase in the size of induration and ulcer. Absence of clinical response: Induration and ulcer area ≤50% compared with the immediately previous evaluation.

Final reports At the end of the study the results will be evaluated and discussed and a final report presented to Colombian army and Ministry of Social Protection, entities sponsoring the project. The relevant results will be published in both, national and international journals, and presented in congresses and scientific meetings.

Ethical aspects This study will be conduced according with the Declaration of Helsinki , the Colombian legislation as per the resolution 008430/93 from the Ministry of Health, Canadian Council of Animal Care, National Institute for drugs and foods vigilance and control - (INVIMA)(Colombia), International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines, and TDR/WHO guidelines for clinical research.

Prior to the admission of the patients in the study, the objectives and the methodology will be explained and informed consent obtained.

The study was approved for the Sede de Investigación Universitaria (SIU) bioethics committee (CBEIH-SIU) and the Leishmaniasis Committee of the Colombian Military Forces.

The right to confidentiality of the patients will be maintained in all the phases of the study.

Competing of interests:

The authors declare that they have no competing of interests.

ELIGIBILITY:
Inclusion Criteria:

* Parasitologically proven cases of CL based on positive smear and/or culture.
* Patients belonging to the National Colombian Army.
* Otherwise healthy subjects on the basis of medical history, physical examination and results of blood test (if seemed necessary by the physician)
* Age 18-40 years.
* Willing to participate in the study, sign the informed consent , to go to the scheduled visits and to the follow-up visits.
* Abstain to receive any other treatment for CL during the trial and follow-up periods.
* Non purulent lesions.
* Mentally sane volunteers.
* No Leishmaniasis treatment in the six months prior to the recruitment.
* Number of lesions no more than 5

Exclusion criteria:

* None of the lesions must be close to the anal, oral and nasal mucosa, or next to the urogenital and anal canal.
* Serious systemic illnesses (as judged by the physician)
* Patients with mucosal compromise.
* Patients with diffuse Leishmaniasis ( defined as 10 or more cutaneous lesions and negative Montenegro's test)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 437 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan D. Vélez, MD. PhD., Principal Investigator — Program for Research and Control in Tropical Diseases - PECET (Director)
Locations (1):
- Program for Research and Control in Tropical Diseases - PECET, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.World Health Organization. Division of Control of Tropical Diseases. Leishmaniasis control home page. [Consultado: 20 de septiembre de 2006]. Disponible en: www.who.int/health-topics/leishmaniasis.htm
- [Background] 2.Echeverry Gaitan MC, Gaona Narváez J, Gualtero SM. Guia de Atención de Leishmaniasis. Revisión y actualización. 2006.
- [Background] Bejarano EE, Uribe S, Rojas W, Dario Velez I. Phlebotomine sand flies (Diptera: Psychodidae) associated with the appearance of urban Leishmaniasis in the city of Sincelejo, Colombia. Mem Inst Oswaldo Cruz. 2002 Jul;97(5):645-7. PMID 12219128
- [Background] Bejarano EE, Uribe S, Rojas W, Velez ID. Presence of Lutzomyia evansi, a vector of American visceral leishmaniasis, in an urban area of the Colombian Caribbean coast. Trans R Soc Trop Med Hyg. 2001 Jan-Feb;95(1):27-8. doi: 10.1016/s0035-9203(01)90320-7. No abstract available. PMID 11280058
- [Background] Agudelo LA, Uribe J, Sierra D, Ruiz F, Velez ID. Presence of American cutaneous Leishmaniasis vectors surrounding the city of Medellin, Colombia. Mem Inst Oswaldo Cruz. 2002 Jul;97(5):641-2. PMID 12219126
- [Background] Berman J. Report to 1999 Miltefosine PDT of the phase II study. 1999. WHO/TDR.
- [Background] Croft SL, Neal RA, Pendergast W, Chan JH. The activity of alkyl phosphorylcholines and related derivatives against Leishmania donovani. Biochem Pharmacol. 1987 Aug 15;36(16):2633-6. doi: 10.1016/0006-2952(87)90543-0. PMID 3606662
- [Background] Ministerio de Proteccion Social, Instituto Nacional de Salud, and SIVIGILA. informe Leishmaniasis semestre 2005. http://www.ins.gov.co/pdf/vcsp/informe_leishmanisis_1sem_2005.pdf. Fecha de acceso: 09/22/06
- [Background] Leandro C, Campino L. Leishmaniasis: efflux pumps and chemoresistance. Int J Antimicrob Agents. 2003 Sep;22(3):352-7. doi: 10.1016/s0924-8579(03)00211-5. PMID 13678842
- [Background] Velez ID, Hendrickx E, Robledo SM, del Pilar Agudelo S. [Gender and cutaneous leishmaniasis in Colombia]. Cad Saude Publica. 2001 Jan-Feb;17(1):171-80. doi: 10.1590/s0102-311x2001000100018. Spanish. PMID 11241940
- [Background] Navin TR, Arana BA, Arana FE, de Merida AM, Castillo AL, Pozuelos JL. Placebo-controlled clinical trial of meglumine antimonate (glucantime) vs. localized controlled heat in the treatment of cutaneous leishmaniasis in Guatemala. Am J Trop Med Hyg. 1990 Jan;42(1):43-50. doi: 10.4269/ajtmh.1990.42.43. PMID 2405727
- [Background] Velasco-Castrejon O, Walton BC, Rivas-Sanchez B, Garcia MF, Lazaro GJ, Hobart O, Roldan S, Floriani-Verdugo J, Munguia-Saldana A, Berzaluce R. Treatment of cutaneous leishmaniasis with localized current field (radio frequency) in Tabasco, Mexico. Am J Trop Med Hyg. 1997 Sep;57(3):309-12. doi: 10.4269/ajtmh.1997.57.309. PMID 9311641
- [Background] Berman JD, Neva FA. Effect of temperature on multiplication of Leishmania amastigotes within human monocyte-derived macrophages in vitro. Am J Trop Med Hyg. 1981 Mar;30(2):318-21. doi: 10.4269/ajtmh.1981.30.318. PMID 7235124
- [Background] Sacks DL, Barral A, Neva FA. Thermosensitivity patterns of Old vs. New World cutaneous strains of Leishmania growing within mouse peritoneal macrophages in vitro. Am J Trop Med Hyg. 1983 Mar;32(2):300-4. doi: 10.4269/ajtmh.1983.32.300. PMID 6837841
- [Background] Neva FA, Petersen EA, Corsey R, Bogaert H, Martinez D. Observations on local heat treatment for cutaneous leishmaniasis. Am J Trop Med Hyg. 1984 Sep;33(5):800-4. doi: 10.4269/ajtmh.1984.33.800. PMID 6091468
- [Background] Wilcocks & Manson-Bahr. Manon's tropical diseases.London: Bailliére Tindall; 1972. p. 119-33.
- [Background] Herwaldt BL, Arana BA, Navin TR. The natural history of cutaneous leishmaniasis in Guatemala. J Infect Dis. 1992 Mar;165(3):518-27. doi: 10.1093/infdis/165.3.518. PMID 1538157
- [Background] Herwaldt BL. Leishmaniasis. Lancet. 1999 Oct 2;354(9185):1191-9. doi: 10.1016/S0140-6736(98)10178-2. PMID 10513726
- [Background] Remme JH, Blas E, Chitsulo L, Desjeux PM, Engers HD, Kanyok TP, Kengeya Kayondo JF, Kioy DW, Kumaraswami V, Lazdins JK, Nunn PP, Oduola A, Ridley RG, Toure YT, Zicker F, Morel CM. Strategic emphases for tropical diseases research: a TDR perspective. Trends Parasitol. 2002 Oct;18(10):421-6. doi: 10.1016/s1471-4922(02)02387-5. PMID 12377584
- [Background] Marsden PD. Mucosal leishmaniasis ("espundia" Escomel, 1911). Trans R Soc Trop Med Hyg. 1986;80(6):859-76. doi: 10.1016/0035-9203(86)90243-9. PMID 3037735
- [Background] Saravia NG, Weigle K, Segura I, Giannini SH, Pacheco R, Labrada LA, Goncalves A. Recurrent lesions in human Leishmania braziliensis infection--reactivation or reinfection? Lancet. 1990 Aug 18;336(8712):398-402. doi: 10.1016/0140-6736(90)91945-7. PMID 1974943
- [Background] Kreutzer RD, Corredor A, Grimaldi G Jr, Grogl M, Rowton ED, Young DG, Morales A, McMahon-Pratt D, Guzman H, Tesh RB. Characterization of Leishmania colombiensis sp. n (Kinetoplastida: Trypanosomatidae), a new parasite infecting humans, animals, and phlebotomine sand flies in Colombia and Panama. Am J Trop Med Hyg. 1991 Jun;44(6):662-75. doi: 10.4269/ajtmh.1991.44.662. PMID 1677544
- [Background] Angulo VM, Tarazona Z, Vega A, Vélez Bernal ID, Betancur Martinez J. Leismaniosis Chagas y Malaria. 27-41. 2002. Colombia, Ascofame.
- [Background] Vélez Bernal ID, Rodriguez Garcia E, Duarte Forero R, López Carvajal L, Castaño Arbeláez M. Enfermedades Tropicales. Guia de manejo de ETV y accidente ofídico. 17-55. 2005. Colombia, PECET
- [Background] Franke ED, Lucas CM, Tovar AA, Kruger JH, De Rivera MV, Wignall FS. Diffuse cutaneous leishmaniasis acquired in Peru. Am J Trop Med Hyg. 1990 Sep;43(3):260-2. doi: 10.4269/ajtmh.1990.43.260. PMID 2221221
- [Background] Hepburn NC, Tidman MJ, Hunter JA. Aminosidine (paromomycin) versus sodium stibogluconate for the treatment of American cutaneous leishmaniasis. Trans R Soc Trop Med Hyg. 1994 Nov-Dec;88(6):700-3. doi: 10.1016/0035-9203(94)90237-2. PMID 7886779
- [Background] Berman JD. Treatment of New World cutaneous and mucosal leishmaniases. Clin Dermatol. 1996 Sep-Oct;14(5):519-22. doi: 10.1016/0738-081x(96)00048-x. PMID 8889330
- [Background] Hendrickx EP, Agudelo SP, Munoz DL, Puerta JA, Velez Bernal ID. Lack of efficacy of mefloquine in the treatment of New World cutaneous leishmaniasis in Colombia. Am J Trop Med Hyg. 1998 Dec;59(6):889-92. doi: 10.4269/ajtmh.1998.59.889. PMID 9886195
- [Background] Navin TR, Arana BA, Arana FE, Berman JD, Chajon JF. Placebo-controlled clinical trial of sodium stibogluconate (Pentostam) versus ketoconazole for treating cutaneous leishmaniasis in Guatemala. J Infect Dis. 1992 Mar;165(3):528-34. doi: 10.1093/infdis/165.3.528. PMID 1311351
- [Background] Franke ED, Wignall FS, Cruz ME, Rosales E, Tovar AA, Lucas CM, Llanos-Cuentas A, Berman JD. Efficacy and toxicity of sodium stibogluconate for mucosal leishmaniasis. Ann Intern Med. 1990 Dec 15;113(12):934-40. doi: 10.7326/0003-4819-113-12-934. PMID 2173461
- [Background] Rojas R, Valderrama L, Valderrama M, Varona MX, Ouellette M, Saravia NG. Resistance to antimony and treatment failure in human Leishmania (Viannia) infection. J Infect Dis. 2006 May 15;193(10):1375-83. doi: 10.1086/503371. Epub 2006 Apr 7. PMID 16619185
- [Background] Kuhlencord A, Maniera T, Eibl H, Unger C. Hexadecylphosphocholine: oral treatment of visceral leishmaniasis in mice. Antimicrob Agents Chemother. 1992 Aug;36(8):1630-4. doi: 10.1128/AAC.36.8.1630. PMID 1329624
- [Background] Hepburn NC, Nolan J, Fenn L, Herd RM, Neilson JM, Sutherland GR, Fox KA. Cardiac effects of sodium stibogluconate: myocardial, electrophysiological and biochemical studies. QJM. 1994 Aug;87(8):465-72. PMID 7922300
- [Background] Croft SL, Coombs GH. Leishmaniasis--current chemotherapy and recent advances in the search for novel drugs. Trends Parasitol. 2003 Nov;19(11):502-8. doi: 10.1016/j.pt.2003.09.008. No abstract available. PMID 14580961
- [Background] Thakur CP, Kumar M, Pandey AK. Comparison of regimes of treatment of antimony-resistant kala-azar patients: a randomized study. Am J Trop Med Hyg. 1991 Oct;45(4):435-41. doi: 10.4269/ajtmh.1991.45.435. PMID 1659239
- [Background] Singh S, Sivakumar R. Challenges and new discoveries in the treatment of leishmaniasis. J Infect Chemother. 2004 Dec;10(6):307-15. doi: 10.1007/s10156-004-0348-9. PMID 15614453
- [Background] Soto-Mancipe J, Grogl M, Berman JD. Evaluation of pentamidine for the treatment of cutaneous leishmaniasis in Colombia. Clin Infect Dis. 1993 Mar;16(3):417-25. doi: 10.1093/clind/16.3.417. PMID 8384011
- [Background] Soto J, Buffet P, Grogl M, Berman J. Successful treatment of Colombian cutaneous leishmaniasis with four injections of pentamidine. Am J Trop Med Hyg. 1994 Jan;50(1):107-11. doi: 10.4269/ajtmh.1994.50.107. PMID 8304565
- [Background] Amato VS, de Paula JG, Imamura R, Amato Neto V, Duarte MI, Boulos MI, Boulos M, Nicodemo AC, de Mendonca JS. [Treatment of american cutaneous leishmaniasis, with lesions in the mucosa, using pentamidine isethionate]. Rev Soc Bras Med Trop. 1996 Sep-Oct;29(5):477-81. doi: 10.1590/s0037-86821996000500011. Portuguese. PMID 8966312
- [Background] Correia D, Macedo VO, Carvalho EM, Barral A, Magalhaes AV, de Abreu MV, Orge ML, Marsden P. [Comparative study of meglumine antimoniate, pentamidine isethionate and aminosidine sulfate in the treatment of primary skin lesions caused by Leishmania (Viannia) braziliensis]. Rev Soc Bras Med Trop. 1996 Sep-Oct;29(5):447-53. doi: 10.1590/s0037-86821996000500007. Portuguese. PMID 8966308
- [Background] Amato V, Amato J, Nicodemo A, Uip D, Amato-Neto V, Duarte M. [Treatment of mucocutaneous leishmaniasis with pentamidine isothionate]. Ann Dermatol Venereol. 1998 Aug;125(8):492-5. French. PMID 9747313
- [Background] Robledo SM, Puerta JA, Munoz DL, Guardo M, Velez ID. [Efficacy and tolerance of pentamidine for treatment of cutaneous leishmaniasis caused by por L. (V) panamensis in Colombia]. Biomedica. 2006 Oct;26 Suppl 1:188-93. Spanish. PMID 17361854
- [Background] de Paula CD, Sampaio JH, Cardoso DR, Sampaio RN. [A comparative study between the efficacy of pentamidine isothionate given in three doses for one week and N-methil-glucamine in a dose of 20mgSbV/day for 20 days to treat cutaneous leishmaniasis]. Rev Soc Bras Med Trop. 2003 May-Jun;36(3):365-71. Epub 2003 Jul 31. Portuguese. PMID 12908038
- [Background] Andersen EM, Cruz-Saldarriaga M, Llanos-Cuentas A, Luz-Cjuno M, Echevarria J, Miranda-Verastegui C, Colina O, Berman JD. Comparison of meglumine antimoniate and pentamidine for peruvian cutaneous leishmaniasis. Am J Trop Med Hyg. 2005 Feb;72(2):133-7. PMID 15741547
- [Background] Lieber-Mbomeyo A, Lipsker D, Milea M, Heid E. [Rhabdomyolysis induced by pentamidine (Pentacarinat) during treatment of cutaneous leishmaniasis: 2 cases]. Ann Dermatol Venereol. 2002 Jan;129(1 Pt 1):50-2. French. PMID 11937930
- [Background] Lightburn E, Morand JJ, Meynard JB, Kraemer P, Chaudier B, Pages F, Garnotel E, Patte JH, Banzet S, Dampierre H, Lepage J, Morillon M, Boutin JP, Hovette P, Chouc C. [Management of American cutaneous leishmaniasis. Outcome apropos of 326 cases treated with high-dose pentamidine isethionate]. Med Trop (Mars). 2003;63(1):35-44. French. PMID 12891748
- [Background] Delobel P, Pradinaud R. Rhabdomyolysis associated with pentamidine isethionate therapy for American cutaneous leishmaniasis. J Antimicrob Chemother. 2003 May;51(5):1319-20. doi: 10.1093/jac/dkg195. Epub 2003 Mar 28. No abstract available. PMID 12668576
- [Background] Hauben M, Reich L. A case report of rhabdomyolysis with pentamidine that prompted a retrospective evaluation of a pharmacovigilance tool under investigation. Br J Clin Pharmacol. 2004 Dec;58(6):675-6. doi: 10.1111/j.1365-2125.2004.02215.x. No abstract available. PMID 15563366
- [Background] Invetigator's Brochure Miltefosine. D-18506. 27-10-1999. Frankfurt, Alemania, ASTA Medica
- [Background] Croft SL, Snowdon D, Yardley V. The activities of four anticancer alkyllysophospholipids against Leishmania donovani, Trypanosoma cruzi and Trypanosoma brucei. J Antimicrob Chemother. 1996 Dec;38(6):1041-7. doi: 10.1093/jac/38.6.1041. PMID 9023651
- [Background] Sundar S, Rosenkaimer F, Makharia MK, Goyal AK, Mandal AK, Voss A, Hilgard P, Murray HW. Trial of oral miltefosine for visceral leishmaniasis. Lancet. 1998 Dec 5;352(9143):1821-3. doi: 10.1016/S0140-6736(98)04367-0. PMID 9851383
- [Background] Verweij J, Planting A, van der Burg M, Stoter G. A dose-finding study of miltefosine (hexadecylphosphocholine) in patients with metastatic solid tumours. J Cancer Res Clin Oncol. 1992;118(8):606-8. doi: 10.1007/BF01211805. PMID 1325463
- [Background] Soto J, Arana BA, Toledo J, Rizzo N, Vega JC, Diaz A, Luz M, Gutierrez P, Arboleda M, Berman JD, Junge K, Engel J, Sindermann H. Miltefosine for new world cutaneous leishmaniasis. Clin Infect Dis. 2004 May 1;38(9):1266-72. doi: 10.1086/383321. Epub 2004 Apr 9. PMID 15127339
- [Background] Alvaro Ruíz Morales, Luis Enrique Morrillo Zárate. Epidemiología clínica. Bogotá, Editorial Médica Panamericana
- [Derived] Lopez L, Cruz C, Godoy G, Robledo SM, Velez ID. Thermotherapy effective and safer than miltefosine in the treatment of cutaneous leishmaniasis in Colombia. Rev Inst Med Trop Sao Paulo. 2013;55(3):S0036-46652013000300197. doi: 10.1590/S0036-46652013000300011. PMID 23740007
- [Derived] Lopez L, Robayo M, Vargas M, Velez ID. Thermotherapy. An alternative for the treatment of American cutaneous leishmaniasis. Trials. 2012 May 17;13:58. doi: 10.1186/1745-6215-13-58. PMID 22594858
- See also: PECET Web Page — http://pecet-colombia.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out between June 2006 and April 2008. The subjects of the study were adult males serving in the Colombian Army. The study was carried out in five military health establishments located in central, northeast and southern Colombia.
Pre-assignment Details: Screening was performed to 486 volunteers, of whom 49 were excluded for several reasons, as follows: Failure to meet inclusion criteria (n=12), unwillingness to participate (n=14) and completion of military service within 6 months (n=23)
Period: Overall Study
Arm/Group | Miltefosine | Glucantime® | Thermotherapy
Started | 145 | 143 | 149
Completed | 121 | 121 | 134
Not Completed | 24 | 22 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miltefosine | Glucantime® | Thermotherapy | Total
Number analyzed (Participants) | 145 | 143 | 149 | 437
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [19 to 37] | 23 [19 to 38] | 23 [19 to 39] | 23 [19 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 145 | 143 | 149 | 437
Region of Enrollment [Number; unit: participants]
  Colombia | 145 | 143 | 149 | 437

OUTCOME MEASURES:

1. Primary Outcome: Complete Clinical Response
Description: Complete Clinical response: Initial cure plus the absence of recurrences or mucosal lesions for 6 months after the end of treatment.
  Note: nitial cure: Complete re-epithelialization of all ulcers and complete disappearance of the induration up to 3 months after the end of treatment.
Time Frame: Until 6 months posttreatment
Population: The efficacy of the treatments was calculated by intention to treat and by protocol.
Measure: Number; unit: participants
Arm/Group | Miltefosine | Glucantime® | Thermotherapy
Number analyzed (Participants) | 145 | 143 | 149
participants | 85 | 103 | 86

2. Secondary Outcome: Recurrence
Description: Reactivation of the lesion at the original site after cure or mucosal compromise during follow-up.
Time Frame: Until 6 months post-treatment
Measure: Number; unit: Participants
Arm/Group | Miltefosine | Glucantime® | Thermotherapy
Number analyzed (Participants) | 145 | 143 | 149
Participants | 3 | 4 | 6

3. Primary Outcome: Failure
Description: At least 50% increase in lesion size at the end of treatment, absence of clinical response at 6 weeks, or any sign of lesion activity 3 months after the end of treatment
Time Frame: Until 3 months posttreatment
Measure: Number; unit: participants
Arm/Group | Miltefosine | Glucantime® | Thermotherapy
Number analyzed (Participants) | 145 | 143 | 149
participants | 34 | 14 | 42

ADVERSE EVENTS:
Time Frame: During treatment and 6 months after treatment
Description: The Risk population differs across Adverse Events terms because not all lab tests were available at all study sites.
Arm/Group | Miltefosine | Glucantime® | Thermotherapy
Serious Adverse Events (participants affected / at risk) | 1/145 | 3/143 | 0/149
Other Adverse Events (participants affected / at risk) | 125/145 | 121/143 | 110/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miltefosine (N=145) | Glucantime® (N=143) | Thermotherapy (N=149)
Death in combat (Social circumstances) | 0 (0) | 2 (2) | 0 (0)
Stab wound (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Miltefosine (N=145) | Glucantime® (N=143) | Thermotherapy (N=149)
Fever (Middle of treatment) (General disorders) | 8/130 (8) | 11/119 (11) | 4/124 (4)
Myalgia (Middle of treatment) (Musculoskeletal and connective tissue disorders) | 9/130 (9) | 12/119 (12) | 3/124 (3)
Arthralgia (Middle of treatment) (Musculoskeletal and connective tissue disorders) | 9/130 (9) | 17/119 (17) | 3/124 (3)
Cephalea (Middle of treatment) (General disorders) | 23/130 (23) | 17/119 (17) | 10/124 (10)
Vomiting (Middle of treatment) (Gastrointestinal disorders) | 29/130 (29) | 3/119 (3) | 3/124 (3)
Nausea (Middle of treatment) (Gastrointestinal disorders) | 38/130 (38) | 4/119 (4) | 5/124 (5)
Anorexia (Middle of treatment) (Gastrointestinal disorders) | 19/130 (19) | 8/119 (8) | 5/124 (5)
BUN (Middle of treatment) (Renal and urinary disorders) | 0/94 (0) | 4/99 (4) | 1/96 (1)
ALT (Middle of treatment) (Hepatobiliary disorders) | 17/132 (17) | 19/137 (19) | 8/106 (8)
Amylase (Middle of treatment) (Hepatobiliary disorders) | 29/112 (29) | 15/111 (15) | 6/87 (6)
Fever (End of treatment) (General disorders) | 8/129 (8) | 29/131 (29) | 4/132 (4)
Myalgia (End of treatment) (Musculoskeletal and connective tissue disorders) | 16/129 (16) | 67/131 (67) | 4/132 (4)
Arthralgia (End of treatment) (Musculoskeletal and connective tissue disorders) | 13/129 (13) | 65/131 (65) | 3/132 (3)
Cephalea (End of treatment) (General disorders) | 30/129 (30) | 52/131 (52) | 13/132 (13)
Vomiting (End of treatment) (Gastrointestinal disorders) | 44/129 (44) | 16/131 (16) | 2/132 (2)
Nausea (End of treatment ) (Gastrointestinal disorders) | 59/129 (59) | 27/131 (27) | 4/132 (4)
Anorexia (End of treatment ) (Gastrointestinal disorders) | 37/129 (37) | 45/131 (45) | 6/132 (6)
Diarrhea (End of treatment) (Gastrointestinal disorders) | 6/129 (6) | 2/131 (2) | 1/132 (1)
Abdominal Pain (End of treatment) (Gastrointestinal disorders) | 9/129 (9) | 2/131 (2) | 0/132 (0)
BUN (End of treatment) (Renal and urinary disorders) | 3/102 (3) | 1/114 (1) | 2/78 (2)
AST (End of treatment) (Hepatobiliary disorders) | 5/103 (5) | 11/111 (11) | 2/75 (2)
ALT (End of treatment) (Hepatobiliary disorders) | 15/92 (15) | 11/90 (11) | 12/105 (12)
Amylase (End of treatment ) (Hepatobiliary disorders) | 11/108 (11) | 24/109 (24) | 7/70 (7)
Haemoglobin (End of treatment) (Blood and lymphatic system disorders) | 1/98 (1) | 7/108 (7) | 2/70 (2)
Creatinine (middle of treatment) (Renal and urinary disorders) | 8/120 (8) | 12/112 (12) | 7/87 (7)
Creatinine (end of treatment) (Renal and urinary disorders) | 6/99 (6) | 1/115 (1) | 1/81 (1)
Lesion pain (middle of treatment) (Skin and subcutaneous tissue disorders) | 14/130 (14) | 3/119 (3) | 27/124 (27)
Lesion infection (middle of treatment) (Skin and subcutaneous tissue disorders) | 5/130 (5) | 2/119 (2) | 9/124 (9)
AST (Middle of treatment) (Hepatobiliary disorders) | 8/105 (8) | 8/99 (8) | 11/93 (11)
Haemoglobin (middle of treatment (Blood and lymphatic system disorders) | 5/113 (5) | 5/107 (5) | 5/96 (5)
Lesion pain (end of treatment) (Skin and subcutaneous tissue disorders) | 11/129 (11) | 16/131 (16) | 18/122 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No